CLINICAL TRIAL: NCT06058663
Title: Phase 1 Trial of Safety and Preliminary Efficacy of Segmental Ablative Radioembolization in Combination With Tremelimumab Plus Durvalumab (MEDI4736) in Patients With Unresectable, or Oligo-Metastatic Cholangiocarcinoma Who Are Not Candidates for Curative Therapy (RAIDEN Trial)
Brief Title: Radioembolization With Tremelimumab and Durvalumab for Locally Advanced Unresectable or Oligo-Metastatic Intrahepatic Cholangiocarcinoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MC1943; NCI-2023-05200 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21-007474 (Other: Mayo Clinic Institutional Review Board); MC1943 (Other: Mayo Clinic)
Record Dates: First submitted 2023-09-06; First posted 2023-09-28 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Locally Advanced Intrahepatic Cholangiocarcinoma; Oligometastatic Intrahepatic Cholangiocarcinoma; Stage III Intrahepatic Cholangiocarcinoma AJCC v8; Stage IV Intrahepatic Cholangiocarcinoma AJCC v8; Unresectable Intrahepatic Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Cerebral Angiography; Biopsy; Specimen Handling; durvalumab; Immunoglobulin G; Disulfides; Magnetic Resonance Spectroscopy; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort I: (Y90, tremelimumab on day 1, cycle 1, durvalumab) (Experimental): Patients receive transarterial Y90 radioembolization and tremelimumab IV over 1 hour on day 1 of cycle 1 and durvalumab IV over 1 hour on day 1 of each cycle. Cycles repeat every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo mapping angiography during screening as well as CT and MRI or PET/CT during screening and on study. Patients also undergo blood sample collection throughout the trial and may undergo tumor biopsy during screening and on study.
  Interventions: Procedure: Angiography; Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Durvalumab; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Biological: Tremelimumab; Procedure: Yttrium-90 Microsphere Radioembolization
- Cohort II: (Y90, tremelimumab on day 14, cycle 1, durvalumab ) (Experimental): Patients receive transarterial Y90 radioembolization on day 1 of cycle 1 and receive tremelimumab IV over 1 hour on day 14 of cycle 1 and durvalumab IV over 1 hour on day 14 of each cycle. Cycles repeat every 42 days for cycle 1 and then every 28 days for cycles 2-24 in the absence of disease progression or unacceptable toxicity. Patients also undergo mapping angiography during screening, as well as CT and MRI or PET/CT during screening and on study. Patients also undergo blood sample collection throughout the trial and may undergo tumor biopsy during screening and on study.
  Interventions: Procedure: Angiography; Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Durvalumab; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Biological: Tremelimumab; Procedure: Yttrium-90 Microsphere Radioembolization

INTERVENTIONS:
Procedure: Angiography — Undergo mapping angiography
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI-4736; MEDI4736
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Biological: Tremelimumab — Given IV
  Other Names: Anti-CTLA4 Human Monoclonal Antibody CP-675,206; CP-675; CP-675,206; CP-675206; Imjudo; Ticilimumab; Tremelimumab-actl
Procedure: Yttrium-90 Microsphere Radioembolization — Receive transarterial Y90 radioembolization
  Other Names: Yttrium Y 90 Microsphere Therapy; Yttrium-90 Radioembolization

SUMMARY:
This phase I trial tests the safety and side effects of yttrium-90 (Y90) radioembolization combined with immunotherapy drugs tremelimumab and durvalumab in treating patients with intrahepatic cholangiocarcinoma (cancer of the bile ducts in the liver) that has spread to nearby tissue or lymph nodes (locally advanced) and cannot be removed by surgery (unresectable) who are not candidates for curative therapy or that has spread from where it first started (primary side) to multiple other places in the body (oligo-metastatic). Cholangiocarcinoma is a rare but aggressive cancer with limited curative options outside of surgery. Immunotherapy has shown modest benefit in hepatobiliary (liver, bile ducts, and gallbladder) cancers including cholangiocarcinoma. Radioembolization is a type of radiation therapy used to treat liver cancer that is advanced or has come back where tiny beads that hold the radioactive substance (radioisotope) yttrium Y90 are injected into or near the hepatic artery (the main blood vessel that carries blood to the liver). The beads collect in the tumor and the Y90 gives off radiation. This destroys the blood vessels that the tumor needs to grow and kills the tumor cells. A monoclonal antibody is a type of protein that can bind to certain targets in the body, such as molecules that cause the body to make an immune response (antigens). Immunotherapy with monoclonal antibodies, such as durvalumab and tremelimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving Y90 radioembolization in combination with tremelimumab and durvalumab immunotherapy may be safe and beneficial in treating patients with locally advanced, unresectable or oligo-metastatic intrahepatic cholangiocarcinoma who are not candidates for curative therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Characterize the safety of the combination of Y90 transarterial radioembolization (TARE), durvalumab and tremelimumab.

SECONDARY OBJECTIVES:

I. Overall efficacy of Y90 + tremelimumab + durvalumab as gauged by response rate (Modified Response Evaluation Criteria in Solid Tumors (mRECIST).

II. Median progression free survival (PFS) and overall survival (OS). III. Infield and out of field objective response rate (complete response and partial response) rate (mRECIST and) in-field and out-of- field duration of response.

IV. Resectability rate. V. Time to respond in treated and non treated lesions.

VI. Correlatives:

VIa. Circulating tumor deoxyribonucleic acid (ctDNA) monitoring per investigator discretion; VIb. Post-treatment dose volume histograms will be obtained using Simplicity software; VIbi. Tissue and blood banking for testing such as immunohistochemistry and Tissue Digital Spatial Profiling - list of biomarkers: CD68, CD 86, CD163, CSF1R - macrophage, M1/M2 markers, CD3 - T-cell differentiator, FoxP3, CD25, CD4 and 8 - T-cell lineage, PD-1, PD-L1, etc. - checkpoints, granzyme B - cytotoxic T lymphocytes (CTL) activity. Next generation (Gen) profiling and ribonucleic acid (RNA) sequencing. Microsatellite instability (MSI)/ mismatch repair (MMR) status, tumor mutational burden (TMB).

EXPLORATORY OBJECTIVES:

I. Tissue and blood for predictive and prognostic biomarkers will be collected.

OUTLINE: Patients are assigned to 1 of 2 arms.

Arm I (COHORT I): Patients receive transarterial Y90 radioembolization and tremelimumab intravenously (IV) over 1 hour on day 1 of cycle 1 and durvalumab IV over 1 hour on day 1 of each cycle. Cycles repeat every 28 days for up to 24 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo mapping angiography during screening as well as computerized tomography (CT) and magnetic resonance imaging (MRI) or positron emission tomography (PET)/CT during screening and on study. Patients also undergo blood sample collection throughout the trial and may undergo tumor biopsy during screening and on study.

Arm II (COHORT II): Patients receive transarterial Y90 radioembolization on day 1 of cycle 1 and receive tremelimumab IV over 1 hour on day 14 of cycle 1 and durvalumab IV over 1 hour on day 14 of each cycle. Cycles repeat every 42 days for cycle 1 and then every 28 days for cycles 2-24 in the absence of disease progression or unacceptable toxicity. Patients also undergo mapping angiography during screening, as well as CT and MRI or PET/CT during screening and on study. Patients also undergo blood sample collection throughout the trial and may undergo tumor biopsy during screening and on study.

Cohort III: This is a dose expansion cohort where patients are enrolled based on the efficacy and safety results from Cohorts I and II.

After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years with body weight > 30 kg
* Histologically or cytologically confirmed, locally advanced intrahepatic cholangiocarcinoma that is not amenable to resection, transplantation, or thermal ablation. Oligometastatic intrahepatic cholangiocarcinoma is also eligible. Specifically, such patients must have EITHER =< 3 malignant extrahepatic lymph nodes (short axis diameter >= 3cm) OR metastatic lesions in one organ other than liver (if only single lesion is present diameter MUST be < 3cm, if up to 3 lesions in one organ each lesion MUST be =< 1cm)
* Measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Hemoglobin >= 9.0 g/dL (=< 14 days prior to registration)
* Absolute neutrophil count (ANC) >= 1000/mm^3 (=< 14 days prior to registration)
* Platelet count >= 75,000/mm^3 (=< 14 days prior to registration)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (patients with known Gilbert disease who have serum bilirubin level 3 x ULN may be enrolled) (=< 14 days prior to registration)
* Alanine aminotransferase (ALT) and aspartate transaminase (AST) =< 5 x ULN (=< 14 days prior to registration)
* Calculated creatinine clearance >= 40 ml/min using the Cockcroft- Gault formula or measured creatinine clearance > 40 ml/min (=< 14 days prior to registration)
* International normalized ratio (INR) =< 1.6. Note: INR prolongation due

  * Anticoagulation (INR >= 2.0 but =< 3.0)) for prophylaxis in patients without liver cirrhosis could be exception
* Adequate hepatic function Child Pugh A and albumin-bilirubin (ALBI) 1 or 2
* Patients with concurrent hepatitis B (HBV) or hepatitis C virus (HCV) infection should meet the following criteria:

  * Patient with HBV or should be monitored for viral levels during study participation
  * Patient with detectable hepatitis B surface antigen (HBsAg) or detectable HBV DNA should have HBV DNA < 100 IU/ml and should be managed per local guidelines
  * Controlled hepatitis B subjects will be allowed if they have started treatment prior to or by the time point of enrollment into the study and treatment is continued during study participation and for >= 6 months after end of study treatment
  * Patients positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Negative urine pregnancy test done prior =< 7 days registration, for persons of childbearing potential only

  * NOTE: If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required

Exclusion Criteria:

* Concurrent enrollment in another clinical study, unless it is an observational clinical study or during the follow up period of an interventional study
* Surgery =< 28 days prior to registration
* Chemotherapy =< 4 weeks prior to registration
* History of > 1 prior systemic therapy for cholangiocarcinoma not including that in the adjuvant setting. Patients who progressed during or =< 6 months from completion of adjuvant therapy are excluded
* Any unresolved toxicity National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) grade >= 2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

  * Patients with grade >= 2 neuropathy will be evaluated on a case-by-case basis after consultation with the study physician
  * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or tremelimumab may be included only after consultation with the study physician
  * History of previous locoregional therapy
  * Previous use of therapeutic cancer vaccines
* Unstable liver function and/ or a change in Child Pugh score during screening

  * Child Pugh B or greater
  * ALBI grade > 2
  * Model for End-Stage Liver Disease (MELD) > 10
* Patient is unable to undergo mapping angiography or mapping angiography demonstrates tumor blood supply that does not lend itself to transarterial therapy
* A lung shunt fraction greater than 30 Gy within a single session, or cumulative does greater than 50Gy
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy

  * NOTE: Patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial
* Active or uncontrolled autoimmune or inflammatory disorders (including Inflammatory bowel disease, systemic lupus erythematosus, rheumatoid arthritis, granulomatosis with polyangiitis, sarcoidosis, Grave's disease)
* History of another primary malignancy except for:

  * Malignancy treated with curative intent and with no known active disease >= 5 years prior to registration and of low potential of recurrence
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing uncontrolled infections including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis (TB) testing in line with local practice), human immunodeficiency virus (HIV), hepatitis B and hepatitis C
  * Serious chronic gastrointestinal condition associated with diarrhea
  * Symptomatic congestive heart failure
  * Unstable angina pectoris, cardiac arrhythmia and uncontrolled hypertension
  * Chronic pulmonary disease including interstitial lung disease requiring oxygen
  * Psychiatric illness/social situations limiting compliance that would limit compliance with study requirement, substantially increase risk of incurring adverse events (AEs) or compromise the ability of the patient to give written informed consent
  * Uncontrolled hypertension
* History of leptomeningeal carcinomatosis
* History of allogeneic transplantation
* Current or prior use of immunosuppressive medication < 14 days before registration. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections
  * Systemic corticosteroids at physiologic doses not to exceed 10mg/day of
  * Prednisone or its equivalent
* Known allergy or hypersensitivity to durvalumab and tremelimumab or any of the constituents of the products
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Pregnant or lactating female
* Life expectancy < 3 months
* Intolerance to contrast agents that is refractory to medical management
* Any other condition which the investigator believes would make participation in the study not acceptable
* History of primary immunodeficiency
* Patients who are unable to consent because they do not understand the nature, significance and implications of the clinical trial and therefore cannot form a rational intention in the light of the facts
* Receipt of live attenuated vaccine < 30 days prior to registration and without need to receive any live attenuated vaccines during study conduct and for up to 30 days after end of durvalumab treatment or 90 days after end of tremelimumab treatment respectively
* Prior immunotherapy such as durvalumab or pembrolizumab is allowed as long as patient does not have progressive disease on it

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) (Cohort 1) | Day 0 to day 28
  Dose-limiting toxicities (DLTs) will be defined as an adverse event (AE) attributed as definitely, probably, or possibility related to the study treatment in the first cycle. All the relevant results pertaining to toxicity will be examined in an exploratory and hypothesis-generating fashion. The number and severity of all adverse events will be tabulated and summarized in this patient population. The grade 3+ AEs will also be described and summarized in a similar fashion. Toxicity is defined as AEs that are classified as either possibly, probably, or definitely related to study treatment. Non-hematologic toxicities will be evaluated via the ordinal Common Terminology Criteria (CTC) standard toxicity grading. Hematologic toxicity measures of thrombocytopenia, neutropenia, and leukopenia will be assessed using continuous variables as the outcome measures (primarily nadir) as well as categorization via CTC standard toxicity grading. Overall toxicity will be explored and summarized.
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) (Cohort 2) | Day 14 to day 42
  DLTs will be defined as an AE attributed as definitely, probably, or possibility related to the study treatment in the first cycle. All the relevant results pertaining to toxicity will be examined in an exploratory and hypothesis-generating fashion. The number and severity of all adverse events will be tabulated and summarized in this patient population. The grade 3+ AEs will also be described and summarized in a similar fashion. Toxicity is defined as AEs that are classified as either possibly, probably, or definitely related to study treatment. Non-hematologic toxicities will be evaluated via the ordinal CTC standard toxicity grading. Hematologic toxicity measures of thrombocytopenia, neutropenia, and leukopenia will be assessed using continuous variables as the outcome measures (primarily nadir) as well as categorization via CTC standard toxicity grading. Overall toxicity will be explored and summarized.

SECONDARY OUTCOMES:
Overall efficacy | Up to 24 months
  Will be assessed by response rate modified Response Evaluation Criteria in Solid Tumors (mRECIST) and Positron Emission Tomography (PET) (PERCIST).
Median progression free survival | Up to 24 months
  Timed endpoints and will be examined in an exploratory and hypothesis-generating fashion.
Median overall survival | Up to 24 months
  Timed endpoints and will be examined in an exploratory and hypothesis-generating fashion.
Objective response rate (complete response and partial response) | From the start of the treatment until disease progression/recurrence, assessed up to 24 months
  Best response is defined to be the best objective status. The modified RECIST version 1.1, mRECIST and PERCIST criteria will be used for tumor evaluation and patients. Responses will be summarized by simple descriptive summary statistics delineating complete and partial responses as well as stable and progressive disease in this patient population (overall and by tumor group).
Duration of response | Up to 24 months
  The modified RECIST version 1.1, mRECIST and PERCIST criteria will be used for tumor evaluation and patients. Responses will be summarized by simple descriptive summary statistics delineating complete and partial responses as well as stable and progressive disease in this patient population (overall and by tumor group).
Change in white blood cell count (WBC) | Up to 24 months
  Assessed by blood test
Change in absolute neutrophil count (ANC) | Up to 24 months
  Assessed by blood test
Change in absolute monocyte count (AMC) | Up to 24 months
  Assessed by blood test
Change in absolute neutrophil count to absolute lymphocyte count (ANC:ALC) ratio | Up to 24 months
  Assessed by blood test
Change in myeloid to lymphoid lineage (M:L) | Up to 24 months
  Assessed by blood test
Change in circulating tumor DNA (ctDNA) | Up to 24 months
  Assessed using Guardant 360 at baseline and throughout treatment
Change in tumor biopsy | Up to 24 months
  Assessed by reviewing pre- and post-biopsies for predictive biomarkers
Change in personalized ctDNA assay | Up to 24 months
  Personalized ctDNA assay recorded and assessed using Signatera bespoke multiplex PCR (mPCR) Next-Generation Sequencing (NGS) assay by Natera, specific to each patient's tumor mutational signatures

CONTACTS AND LOCATIONS:
Overall Officials: Umair Majeed, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials